CLINICAL TRIAL: NCT04183426
Title: Tonometry(1) and Duplex Ultrasound(2) to Predict Cardiovascular Events in to be Treated Patients With an Abdominal Aortic Aneurysm (One-Two-Treat Trial)
Brief Title: Tonometry(1) and Duplex Ultrasound(2) to Predict CV Events in to be Treated Patients With an AAA
Acronym: One-Two-Treat
Status: Recruiting | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Radboud University Medical Center (Other); Canisius-Wilhelmina Hospital (Other); Gelderse Vallei Hospital (Other); Medisch Spectrum Twente (Other); Deventer Ziekenhuis (Other); Gelre Hospitals (Other); Maxima Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: One-Two-Treat Trial
Record Dates: First submitted 2019-11-19; First posted 2019-12-03 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Aortic Aneurysm; Cardiovascular Events
Keywords: Functional Response; Abdominal Aortic Aneurysm; Cardiovascular Events
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Vascular Stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Carotid Artery Reactivity test (CAR test) — The CAR test will be applied to stimulate the sympathetic nervous system. This thermal stimulus is known to elevate blood pressure via sympathetic pathways, so it can be used to study the vascular response to sympathetic activation. The participant will submerge their left hand in a bucket of ice water (approximately 4 degrees celcius) for 3 minutes, which is reported to be sufficient to induce a maximal dilation in the common carotid artery. At baseline and every minute after the hand is submerged in ice water, the blood pressure will be measured to check whether a sympathetic stimulation is achieved.
Diagnostic Test: Arterial Stiffness — The SphygmoCor device will be used to non-invasively measure arterial stiffness parameters using applanation tonometry. For Pulse Wave Analyses (PWA), the radial waveform will be recorded. Approximately 10 waveforms are averaged, resulting in several non-invasive parameters:
  * Peripheral pressure parameters
  * Central and abdominal aneurysm pressure parameters (derived using a transfer function)
  * Cardiac output parameters (sub-endocardial viability ratio (SEVR), Ejection Duration (ED))
  Pulse wave velocity will be performed by recording the waveforms of the carotid and femoral artery sequentially. The travelled distance will be measured according to the current guidelines and entered in the program. The program will calculate the PWV based on 10 ECG triggered waveform of each artery.

SUMMARY:
Abdominal aortic aneurysm (AAA) is a common vascular disease and associated with risk of rupture, but also with a high cardiovascular (CV) event rate. A key difficulty in AAA is predicting these life-threatening complications, which are strongly linked to vascular health. In 2013, the SMART risk score was developed to calculate the risk of the patients for recurrent vascular events based on clinical characteristics. Recently, a novel, easy to perform, non-invasive test of endothelial function (the carotid artery reactivity (CAR) test), reflecting target organ damage, has been introduced. The CAR is a simple, quick (5-min), non-invasive test that uses ultrasound to examine the carotid artery in response to sympathetic stimulation by placing one hand in cold water. This test shows strong agreement with both coronary and aortic responses to sympathetic stimulation and predicted CV-events in patients with peripheral arterial disease.

The aim of this prospective 2-year follow-up study is to investigate the predictive capacity of the CAR-test for development of CV-events after elective AAA repair in comparison to the SMART risk score. Secondary objectives are to investigate the predictive capacity of arterial stiffness measurements and the post-operative CAR-test for development of CV-events and to evaluate health status scores to provide insight if these scores can support clinical decision making.

DETAILED DESCRIPTION:
The investigators will include 194 patients with an AAA who will be scheduled for repair. Participants will be recruited from all collaborating hospitals (currently Radboudumc, Rijnstate, CWZ) after providing written informed consent.

In this observational, prospective study, a total of 194 patients who are going to be treated for their AAA will be included. Baseline patient characteristics will be registered, including traditional risk factors and CV-history. In addition to regular care of measuring AAA diameter progression (in mm/year), we will perform the CAR-test (10-min) and non-invasive arterial stiffness measures (PWA and PWV) with the SphygmoCor device (10-min).

Furthermore, the investigators will ask patients to complete a questionnaire about the quality of their life. A second questionnaire tries to clarify the disease experience of the patients. Both questionnaires will be asked to be completed at the start, 6-8 weeks after repair, after one year and after two years of repair. Subsequently, the investigators will record major adverse cardiovascular events (MACE) according to the International Classification of Disease-10. Registration of MACE will be performed using hospital-records and following international guidelines. Across a 2-year follow-up, by means of regular follow-up appointments, the investigators will examine the ability of the CAR parameter and arterial stiffness parameters to predict CV-events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old;
* Informed consent form understood and signed and patient agrees to follow- up visits;
* Has an infrarenal or juxtarenal abdominal aortic aneurysm (AAA), scheduled for elective repair (i.e open repair, EVAR, FEVAR and CHEVAR) according to standard practice;

Exclusion Criteria:

* Life expectancy < 2 years;
* Psychiatric or other condition that may interfere with the study;
* Participating in another clinical study, interfering on outcomes;
* Increased risk for coronary spasms (score Rose-questionnaire ≥2;
* Presence of Raynaud's phenomenon, Marfan syndrome, chronic pain syndrome at upper extremity(s), presence of an AV fistula or shunt, open wounds to the upper extremity(s), and/or scleroderma associated with placing the hand in ice water;
* Recent (<3 months) presence of angina pectoris, myocardial infarction, cerebral infarction, and/or heart failure, or PAD treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an AAA who will be scheduled for repair, will be included. AAA patients will be recruited from all collaborating hospitals (Radboudumc, Rijnstate, CWZ), who provide written informed consent. Additionally, also AAA-patients under surveillance of general practitioners are eligible (and will be contacted through the hospital-links), since the nature of the tests allow for performing all tests at the general practitioners' office.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 2-year follow-up
  Incidence of MACE, including myocardial infarction, cerebral infarction, heart failure, rupture, and peripheral vascular disease

SECONDARY OUTCOMES:
SMART Risk score | Baseline
  Second Manifestations of ARTerial disease risk score is developed to determine the risk of recurrent vascular events based on clinical characteristics of the patients
CAR-test results | Baseline and 6-weeks after operation
  Percentage of vasodilation/vasoconstriction to the CAR test at the common carotid artery at baseline
CAR-test results | Baseline and 6-weeks after operation
  Magnitude of the blood flow and perfusion response
CAR-test results | Baseline and 6-weeks after operation
  Timing of the blood flow and perfusion response
CAR-test results | Baseline and 6-weeks after operation
  Blood pressure responses
CAR-test results | Baseline and 6-weeks after operation
  Heart rate responses
CAR-test results | Baseline and 6-weeks after operation
  Changes after treatment
SphygmoCor parameters | Baseline, 6-weeks, 1 year and 2 year after operation
  Peripheral pressure measurements (PWA)
SphygmoCor parameters | Baseline, 6-weeks, 1 year and 2 year after operation
  Central pressure measurements (derived using a transfer function, PWA)
SphygmoCor parameters | Baseline, 6-weeks, 1 year and 2 year after operation
  Abdominal pressure measurements (derived using a transfer function, PWA)
SphygmoCor parameters | Baseline, 6-weeks, 1 year and 2 year after operation
  SEVR
SphygmoCor parameters | Baseline, 6-weeks, 1 year and 2 year after operation
  ED
SphygmoCor parameters | Baseline, 6-weeks, 1 year and 2 year after operation
  PWV
SphygmoCor parameters | Baseline and 6-weeks after operation
  Change in Peripheral pressure measurements (PWA) after treatment
SphygmoCor parameters | Baseline and 6-weeks after operation
  Change in Central pressure measurements (derived using a transfer function, PWA) after treatment
SphygmoCor parameters | Baseline and 6-weeks after operation
  Change in Abdominal pressure measurements (derived using a transfer function, PWA) after treatment
SphygmoCor parameters | Baseline and 6-weeks after operation
  Change in SEVR after treatment
SphygmoCor parameters | Baseline and 6-weeks after operation
  Change in ED after treatment
SphygmoCor parameters | Baseline and 6-weeks after operation
  Change in PWV after treatment
Score EQ-5D questionnaire | Baseline, 6-weeks, 1 year and 2 year after operation
  Patient reported outcomes measured by the general health questionnaire
Score IPQ-K questionnaire | Baseline, 6-weeks, 1 year and 2 year after operation
  Patient reported outcomes measured by the disease perception questionnaire

OTHER OUTCOMES:
Demographic characteristics | Baseline
  Age
Demographic characteristics | Baseline
  Gender
Demographic characteristics | Baseline
  If current smoker
Demographic characteristics | Baseline
  Height
Demographic characteristics | Baseline
  Weight
Demographic characteristics | Baseline
  ASA class
Demographic characteristics | Baseline
  Medical history
Demographic characteristics | Baseline
  Blood pressure
Demographic characteristics | Baseline
  Heart rate
Demographic characteristics | Baseline
  Cardiac measurements
Demographic characteristics | Baseline
  SVS class
Preoperative anatomic characteristics before primary repair procedure | Baseline
  AAA sac diameter
Preoperative anatomic characteristics before primary repair procedure | Baseline
  Infrarenal aortic neck lumen diameter
Preoperative anatomic characteristics before primary repair procedure | Baseline
  Proximal non-aneurysmal aortic neck length
Preoperative anatomic characteristics before primary repair procedure | Baseline
  Proximal aortic neck angle
Preoperative anatomic characteristics before primary repair procedure | Baseline
  Aneurysm blood lumen diameter
Preoperative anatomic characteristics before primary repair procedure | Baseline
  Common iliac artery diameters
Preoperative anatomic characteristics before primary repair procedure | Baseline
  Blood lumen diameter
Procedure and discharge details of intervention | At time of procedure
  Type of procedure
Procedure and discharge details of intervention | At time of procedure
  Anesthesia type
Procedure and discharge details of intervention | At time of procedure
  Access type
Procedure and discharge details of intervention | At time of procedure
  Used stent lengths
Procedure and discharge details of intervention | At time of procedure
  Contrast volume used
Procedure and discharge details of intervention | At time of procedure
  Total procedure time
Procedure and discharge details of intervention | At time of procedure
  Immediate procedural technical success
Procedure and discharge details of intervention | During procedure
  Complications pre procedure
Procedure and discharge details of intervention | Up to 2 years
  Complications post procedure
Procedure and discharge details of intervention | During procedure
  Additional procedures estimated blood loss
Procedure and discharge details of intervention | During procedure
  Blood transfusion
Procedure and discharge details of intervention | Up to 2 years
  Concomitant procedures
Procedure and discharge details of intervention | After procedure till discharge
  Time in ICU
Procedure and discharge details of intervention | After procedure till discharge
  Time to hospital discharge
Medications | During 2-year follow up
  Dose of Anti-platelets
Medications | During 2-year follow up
  Dose of Anti-coagulants
Medications | During 2-year follow up
  Dose of Anti-hypertensives
Medications | During 2-year follow up
  Dose of Statins
Medications | During 2-year follow up
  Dose of Beta-blockers
Medications | During 2-year follow up
  Dose of Sympathicomimetics
Laboratory test results | 2-year follow-up
  Hemoglobin
Laboratory test results | 2-year follow-up
  Serum creatinine
Laboratory test results | 2-year follow-up
  Cholesterol
Laboratory test results | 2-year follow-up
  eGFR
Laboratory test results | 2-year follow-up
  CRP
Parameters during follow-up | 2-year follow-up
  Any type of endoleak
Parameters during follow-up | 2-year follow-up
  AAA sac expansion
Parameters during follow-up | 2-year follow-up
  Any other (S)AE

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, MD, prof, Principal Investigator — Rijnstate Hospital
Locations (7):
- Netherlands (7):
  - Radboudumc, Nijmegen, Gelderland
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Gelre Hospitals, Apeldoorn
  - Deventer Hospital, Deventer
  - Ziekenhuis Gelderse Vallei, Ede
  - Medisch Spectrum Twente, Enschede
  - Maxima Medical Center, Veldhoven